CLINICAL TRIAL: NCT03278912
Title: Natural History of Intestinal Inflammation in Patients With Primary Immune Dysregulations
Brief Title: Natural History of Intestinal Inflammation in People With Primary Immune Dysregulations
Status: Withdrawn | Type: Observational
Why Stopped: Funding completed.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 170163; 17-I-0163
Record Dates: First submitted 2017-09-09; First posted 2017-09-12 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Chronic Granulomatous Disease; Inflammatory Bowel Disease
Keywords: Inflammatory Bowel Disease; Chronic Granulomatous Disease; Dysbiosis; Microbiome; Immunodeficiency; Natural History
MeSH Terms: conditions — Granulomatous Disease, Chronic; Inflammatory Bowel Diseases; Dysbiosis; Immunologic Deficiency Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- IBD: -Patients with IBD without a diagnosed PIDD.-First- or second-degree relatives of patients with a PIDD of interest who do not have a PIDD themselves, but have diagnosed or suspected IBD.
- Non-PIDD/non-IBD (healthy volunteers): healthy volunteers
- PIDD: CGD cohort; IPEX syndrome cohort; CTLA4 haploinsufficiency cohort; LRBA deficiency and hypomorphic RAG deficiency cohorts

SUMMARY:
Background:

PIDD stands for primary immune dysregulation. It is a general term that includes many different inherited immune system disorders. The immune system is the part of the body that helps fight disease and infection. People with PIDDs can develop many kinds of health problems. One of these is inflammatory bowel disease (IBD), which causes diarrhea and cramping. Researchers want to learn more about these disorders to develop possible treatments.

Objective:

To learn more about when and why IBD may develop in some people with PIDDs.

Eligibility:

People ages 3 and older who have PIDD or IBD.

Healthy volunteers in this age group are also needed.

Design:

Visit 1: Participants will be screened with physical exam, medical history, and blood and urine tests.

Visit 2: Participants will:

* Have more physical exams and blood and urine tests.
* Answer questions about quality of life and food history.
* Provide a stool sample.
* Have nasal and rectal skin swabs.
* Have saliva collected.

Participants will have 1 follow-up visit per year. They will repeat visit 2 procedures.

Participants will be contacted by phone or email in between yearly visits. They will be asked about their health. They will complete a quality-of-life questionnaire and send a stool sample that is collected at home.

If participants experience a sudden change in symptoms or undergo a new treatment, they may be asked to complete visit 2 procedures.

If participants are not able to come to NIH, study data and samples can be collected without an in-person visit.

Participants will have a final study visit about 10 years after Visit 1. They will repeat visit 2 procedures.

DETAILED DESCRIPTION:
Over 1 million people suffer from IBD in the United States. Although the exact pathogenesis is unclear, IBD results from an inappropriate inflammatory response to intestinal microbes which is influenced by the environment in a genetically susceptible host. IBDs can be classified as conventional (Crohn disease (CD) and ulcerative colitis (UC)) and unclassified (early onset, difficult to treat, associated with monogenic disorders and PIDDs). Among the 200 IBD susceptibility loci identified in genome-wide association studies (GWAS), overlap with aberrations identified in PIDDs has been observed, thereby supporting the study of PIDDs to better understand conventional IBD pathogenesis, while recognizing PIDD-associated IBDs as distinct disease entities requiring specialized management.

The prevalence of PIDDs worldwide is estimated at 1 in 2000 live births and encompasses a growing list of over 300 PIDDs. Despite the fact that GI disease is the second most common complication in patients with PIDDs (rates ranging from 5-50%), little is known about PIDDspecific

IBD pathogenesis and even less is understood about the role of the microbiota both as a consequence and modulator of immune response in these inherited disorders. Moreover, there may be a time-limited period ("immunological window of opportunity"), coinciding with the maturation of the host s microbiome, during which early immune education may have long-term effects on predisposition to aberrant immune responses and inflammatory dysregulation. The primary objective of this study is to determine if PIDDs result in intestinal dysbioses, which alter local and systemic immune responses. Our long-term goal is to comprehensively investigate the immunological window of opportunity as it relates to PIDD-associated IBDs to define time-sensitive immunoregulatory targets for therapeutic intervention. We will pursue this goal through a prospective, longitudinal study of pediatric and adult patients with PIDDs (with and without IBD) before and after treatment and/or diagnostic interventions, including but not limited to hematopoietic stem cell transplantation (HSCT). Findings from subjects with PIDDs will be compared to those from subjects with IBD as well as healthy volunteers. This multifaceted study will complement primary patient protocols while allowing for the direct interrogation of specific arms of innate and adaptive immunity in the context of host-microbiome interactions. Patients will be studied over time through the collection of clinical metadata, blood, stool, urine, saliva, skin swabs, and biopsies obtained from clinically-indicated endoscopies in age-appropriate patients. PIDDs of interest include but are not limited to: CGD, CTLA4 and LRBA protein deficiency, hypomorphic RAG deficiency, and IPEX syndrome.

ELIGIBILITY:
* INCLUSION CRITERIA:
* General Inclusion Criteria - All individuals must meet the following criteria to be eligible for study participation:

  * Age greater than or equal to 3 years.
  * Willing to allow storage of samples for future research.
  * Willing to allow genetic testing of their samples.
  * Negative urine or serum pregnancy test for women of childbearing potential.
* Specific Inclusion Criteria for PIDD of Interest Cohort: Enrollment as a patient with confirmed PIDD or carrier status in a current NIH protocol, regardless of an IBD component.
* Specific Inclusion Criteria for IBD Cohort:

  * Enrollment as a patient with confirmed IBD in a current NIH protocol.
  * Absence of clinical findings or history suggestive of a primary or acquired immunodeficiency (not including immunodeficiency caused by certain IBD treatments).
* Specific Inclusion Criteria for non-PIDD/non-IBD Cohort (Healthy Volunteers):

  * Absence of clinical findings or history suggestive of a primary or acquired immunodeficiency.
  * Absence of clinical findings or history suggestive of IBD.

EXCLUSION CRITERIA:

* General Exclusion Criteria - An individual who meets any of the following criteria will be excluded from study participation:

  * Active malignancy requiring treatment.
  * HIV.
  * Current treatment for hepatitis B.
  * Current treatment for hepatitis C.
  * Recreational IV drug use within the past 6 months (based on subject report).
  * Participation in a research study of an investigational vaccine within the past 6 months.
  * Any condition that, in the opinion of the investigator, contraindicates participation in this study.
* Specific Exclusion Criteria for PIDD of Interest Cohort: None.
* Specific Exclusion Criteria for IBD Cohort: None.
* Specific Exclusion Criteria for non-PIDD/non-IBD Cohort (Healthy Volunteers):

  * Treatment with systemic antimicrobials within the past 3 months, unless it is a prophylactic regimen consisting of either an azole , trimethoprim-sulfamethoxazole, a quinolone, or any antimicrobial regimen resembling a typical prophylaxis regimen used to treat a PIDD of interest.
  * Treatment with immune modulators within the past 6 months.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include patients and healthy volunteers greater than or equal to 3 years of age; PIDDs of interest, IBD, and Non-PIDD/non-IBD (healthy volunteers)@@@@@@
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2023-09-08 (Actual)

PRIMARY OUTCOMES:
Disease-specific intestinal microbiome signatures, and related localized and systemic immune responses. | Baseline and Annual follow-up visits spanning 10 years
  1. Microbiome, metabolomics, and transcriptomic signatures will be examined between comparison groups.

SECONDARY OUTCOMES:
Changes in microbiome signatures. Changes in metabolomic and transcriptomic signatures. | Baseline and Annual follow-up visits spanning 10 years
  1. Microbiome, metabolomics, and transcriptomic signatures will be examined between comparison groups.
Changes in systemic and tissue-specific markers of innate and adaptive immunity. | Baseline and Annual follow-up visits spanning 10 years
  2. For evaluation of markers of innate and adaptive immunity (local and systemic) most comparisons will be made using 2-tailed Student t tests with statistical significance set at a p less than or equal to 0.05.
Disease-specific differences in relative quantity and function of peripheral blood and tissue immune cells (includes hematopoietic and stromal cells). | Throughout length of study
  3. For evaluation of disease-specific differences in relative quantity and function of peripheral blood and tissue immune cells most comparisons will be made using 2-tailed Student t tests with statistical significance set at a p less than or equal to 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Christa S Zerbe, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
.The following will be shared:@@@@@@ (Summation)De-identified data in an NIH-funded or approved public repository.@@@@@@ (Summation)Identified data in the Biomedical Translational Research Information System (BTRIS).@@@@@@.De-identified or identified data with approved NIH-based and/or outside collaborators under appropriate agreements.
Supporting Information: SAP
Time Frame: Data will be shared before publication, at publication or shortly after publication.
Access Criteria: Data will be shared through:@@@@@@ (Summation)An NIH-funded or approved public repository: National Center for Biotechnology Information Sequence Read Archive (NCBI SRA) Database.@@@@@@ (Summation)BTRIS.@@@@@@ (Summation)Approved outside collaborators under appropriate individual agreements.@@@@@@ (Summation)Publication and/or public presentations.@@@@@@The PI will review and approve/disapprove requests for IDP.

REFERENCES:
- [Background] Agarwal S, Mayer L. Gastrointestinal manifestations in primary immune disorders. Inflamm Bowel Dis. 2010 Apr;16(4):703-11. doi: 10.1002/ibd.21040. PMID 19637385
- [Background] Marciano BE, Rosenzweig SD, Kleiner DE, Anderson VL, Darnell DN, Anaya-O'Brien S, Hilligoss DM, Malech HL, Gallin JI, Holland SM. Gastrointestinal involvement in chronic granulomatous disease. Pediatrics. 2004 Aug;114(2):462-8. doi: 10.1542/peds.114.2.462. PMID 15286231
- [Background] Uhlig HH. Monogenic diseases associated with intestinal inflammation: implications for the understanding of inflammatory bowel disease. Gut. 2013 Dec;62(12):1795-805. doi: 10.1136/gutjnl-2012-303956. PMID 24203055
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2017-I-0163.html